CLINICAL TRIAL: NCT07139236
Title: Preoperative Endoscopic Ultrasound Elastography for Prediction of Intraoperative Pancreatic Texture and Postoperative Pancreatic Fistula After Pancreaticoduodenectomy: A Prospective Study
Brief Title: Preoperative EUS Elastography for Pancreatic Texture and POPF Prediction After PD
Acronym: EUS-E
Status: Recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Other Study IDs: 1378/12/2024
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Neoplasms; Pancreatic Fistula
Keywords: Pancreatic cancer; EUS; Whipple procedure; EUS-E; Pancreatic surgery; Pancreas; Elastography
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Preoperative Endoscopic Ultrasound Elastography (EUS Elastography): Patients undergoing elective pancreaticoduodenectomy (PD) who will receive preoperative endoscopic ultrasound elastography (EUS elastography) evaluation.
  Interventions: Procedure: Preoperative Endoscopic Ultrasound Elastography (EUS Elastography)

INTERVENTIONS:
Procedure: Preoperative Endoscopic Ultrasound Elastography (EUS Elastography) — All enrolled patients will undergo a preoperative EUS-E examination within one weeks prior to pancreaticoduodenectomy. The EUS-E will be performed by experienced endosonographers using a radial or linear array echoendoscope connected to a compatible ultrasound processor. Both qualitative (color mapping) and quantitative (strain ratio, strain histogram) data will be obtained. Multiple measurements of the strain ratio will be taken from a region of interest within the pancreatic parenchyma adjacent to the lesion. The mean strain ratio will be recorded for analysis. Standard EUS imaging will also be recorded.
  Standard pancreaticoduodenectomy will be performed . Intraoperative pancreatic texture will be subjectively assessed by the surgeon and recorded. Postoperative monitoring for pancreatic fistula will follow established clinical guidelines.

SUMMARY:
This prospective study evaluates whether preoperative endoscopic ultrasound elastography (EUS-E) can predict pancreatic texture during surgery and risk of postoperative pancreatic fistula (POPF) in 100 patients undergoing pancreaticoduodenectomy. EUS-E measures pancreatic stiffness preoperatively. Intraoperative texture ("soft" or "hard") is assessed by surgeons blinded to EUS-E results. POPF is graded using ISGPF criteria. Predictive accuracy of EUS-E will be analyzed statistically.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy is a complex surgery with significant morbidity, primarily due to postoperative pancreatic fistula (POPF). Soft pancreatic texture is a major risk factor for POPF. Endoscopic ultrasound elastography (EUS-E) is a promising tool for assessing tissue stiffness. This study will prospectively enroll patients undergoing PD. Preoperative EUS-E will be performed, and intraoperative pancreatic texture will be assessed by the surgeon. Postoperative outcomes, especially POPF, will be meticulously recorded. The study will analyze the diagnostic accuracy of EUS-E for pancreatic texture, its correlation with POPF severity,, as well as the impact on patient outcomes. Data will be collected from medical records, EUS reports, surgical notes, and pathology reports, with strict quality control and confidentiality measures. Statistical analysis will include Receiver Operating Characteristic (ROC) curve analysis for accuracy, and regression analyses to identify predictors and assess impact on outcomes.

In this study, blinding (masking) is implemented as follows:

* Surgeons are blinded to the results of the preoperative endoscopic ultrasound (EUS) elastography. They do not have access to the pancreatic stiffness measurements before or during surgery, ensuring their intraoperative assessment of pancreatic texture remains unbiased.
* Outcome assessors-those evaluating postoperative pancreatic fistula (POPF) and other clinical outcomes-are also blinded to both the preoperative elastography results and the intraoperative texture assessment. This reduces the risk of detection bias when determining study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Patients scheduled for elective pancreaticoduodenectomy (PD) due to pancreatic head or periampullary disease, including but not limited to:

  * Pancreatic cancer (all stages eligible if resectable)
  * Periampullary cancer
  * Bile duct cancer
  * Duodenal cancer
* Patients deemed suitable for PD by the multidisciplinary pancreatic surgery team based on preoperative imaging and clinical evaluation.
* Adequate organ function and physiological reserve to undergo major abdominal surgery, as determined by clinical assessment and anesthesiology evaluation.

  * Ability to provide written informed consent and comply with study procedures.

Exclusion Criteria:

* Evidence of distant metastases or locally advanced unresectable disease on preoperative imaging or clinical evaluation (e.g., liver metastases, peritoneal carcinomatosis, involvement of major vessels beyond resectability).
* Previous pancreatic surgery or total pancreatectomy.
* Chronic pancreatitis confirmed by clinical, radiological, or histological criteria that could confound pancreatic stiffness assessment.
* Severe comorbidities or American Society of Anesthesiologists (ASA) physical status classification IV or higher, making the patient unfit for surgery.
* Preoperative serum albumin less than 2.5 g/dL, indicating severe malnutrition.
* Patients undergoing neoadjuvant chemotherapy or radiotherapy prior to surgery.
* Pregnancy or lactation.
* Contraindications to EUS (e.g., esophageal obstruction)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults aged 18 and older scheduled for elective pancreaticoduodenectomy (PD) for resectable pancreatic head or periampullary diseases, such as pancreatic cancer, periampullary cancer, distal bile duct cancer and duodenal cancer. Patients must be medically fit for major surgery, with adequate organ function and physiological reserve, based on clinical and anesthesiology assessments. Exclusions apply to those with distant metastases, locally advanced unresectable tumors, prior pancreatic surgery, or chronic pancreatitis to avoid confounding tissue assessment. Patients often present with symptoms like jaundice or abdominal discomfort and are managed in specialized pancreatic centers with multidisciplinary care. This cohort is appropriate for evaluating preoperative endoscopic ultrasound elastography as a tool to predict intraoperative pancreatic texture and postoperative pancreatic fistula risk.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of preoperative EUS elastography in predicting intraoperative pancreatic texture (soft vs. hard). | Intraoperative at the time of pancreaticoduodenectomy (for tactile assessment) and pre-operative (for EUS-E).
  Assessed by calculating sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and overall accuracy of EUS-E parameters (e.g., strain ratio) against the intraoperative tactile assessment of pancreatic texture.

SECONDARY OUTCOMES:
Incidence of Postoperative Pancreatic Fistula (POPF) | Up to 30 days post-surgery.
  Occurrence of POPF classified by the International Study Group on Pancreatic Fistula (ISGPF) grading system (Grades A, B, and C) within 30 days after pancreaticoduodenectomy.
Correlation between EUS Elastography Parameters and POPF Severity. | Preoperative (EUS-E) and postoperative (POPF) evaluated within 30 days post-surgery.
  Relationship between quantitative EUS-E parameters and the incidence and severity of POPF.

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital / Minia university, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No